CLINICAL TRIAL: NCT00005691
Title: Psychosocial Risk Factors for Coronary Heart Disease in Swedish Women
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4213; R01HL045785 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2001-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease

SUMMARY:
To study psychosocial risk factors for coronary heart disease in Swedish women.

DETAILED DESCRIPTION:
BACKGROUND:

The incidence of non-fatal myocardial infarction in Swedish women below age 60 increased during the past 20 years. Standard risk factor change includes a decrease in average systolic blood pressure and S-cholesterol but a moderate increase in smoking and diabetes prevalence. During the same time period Swedish women have 'moved' into the labor market, so that employment rates are now similar in Swedish men and women. However, women have kept the main responsibilities for household and child care. In spite of generous legislation for maternity leave and child care, the strains from multiple roles and responsibilities have probably increased in Swedish women. The study sought to provide an answer to: 1) which factors - biological and behavioral - influenced both the extent of and progress of coronary artery disease, 2) which physiological, biochemical, or neuroendocrine mechanisms participated in the process. In addition to conventional statistical methods, canonical correlations analyses were used to describe direct and indirect pathways of the pathogenesis. Furthermore, by means of the two comparison groups, information was obtained about the specific characteristics of the female psychosocial and behavioral coronary heart disease risk profile.

DESIGN NARRATIVE:

The role of social strain was studied within a broader psychosocial context including social networks, social supports, social skills, reciprocity, coping, stressors, chronic work strain, family structure, personality and behavior characteristics. These aspects were related to possible physiologic cardiovascular mechanisms including reactivity of and persistent elevated heart rates and blood pressure on ambulatory monitoring as well as cardiac dysrhythmia and silent or symptomatic ischemia. Psychoneuroendocrine pathways were also investigated. These included catecholamines, cortisol, prolactin, estrogen, testosterone, gastrin, somatostatin. Other biochemical measures included lipid profile, coagulation, thrombolysis and immune function. These examinations were applied to all women below age 60, living in the greater Stockholm area, with signs or symptoms of coronary heart disease. The women were followed and reexamined (including angiograms) after 2 to 2.5 years. They were compared to an equal number of age matched men and to an equal number of age matched healthy women from the same catchment area.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-09; Study Completion 1996-08 (Actual)

REFERENCES:
- [Background] Horsten M, Wamala SP, Vingerhoets A, Orth-Gomer K. Depressive symptoms, social support, and lipid profile in healthy middle-aged women. Psychosom Med. 1997 Sep-Oct;59(5):521-8. doi: 10.1097/00006842-199709000-00009. PMID 9316185
- [Background] Wamala SP, Wolk A, Orth-Gomer K. Determinants of obesity in relation to socioeconomic status among middle-aged Swedish women. Prev Med. 1997 Sep-Oct;26(5 Pt 1):734-44. doi: 10.1006/pmed.1997.0199. PMID 9327484
- [Background] Wamala SP, Wolk A, Schenck-Gustafsson K, Orth-Gomer K. Lipid profile and socioeconomic status in healthy middle aged women in Sweden. J Epidemiol Community Health. 1997 Aug;51(4):400-7. doi: 10.1136/jech.51.4.400. PMID 9328547
- [Background] Orth-Gomer K, Mittleman MA, Schenck-Gustafsson K, Wamala SP, Eriksson M, Belkic K, Kirkeeide R, Svane B, Ryden L. Lipoprotein(a) as a determinant of coronary heart disease in young women. Circulation. 1997 Jan 21;95(2):329-34. doi: 10.1161/01.cir.95.2.329. PMID 9008445